CLINICAL TRIAL: NCT02104141
Title: An Open Label, Multicenter, Clinical Study of the Safety and Efficacy of the LDR Spine ROI-A Interbody Fusion System Using the VerteBRIDGE™ Plating System
Brief Title: Retrospective/Prospective Data Collection on the LDR ROIA Interbody Fusion Device With VerteBRIDGE Plating
Status: Completed | Type: Observational
Sponsor: LDR Spine USA (Industry)
Responsible Party: Sponsor
Other Study IDs: ROIA100
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Degenerative Disc Disease
Keywords: DDD; lumbar spine; fusion rate; degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Operated Subjects: ROIA Interbody Cage with VerteBRIDGE plating
  Interventions: Device: ROIA Interbody Cage with VerteBRIDGE plating

INTERVENTIONS:
Device: ROIA Interbody Cage with VerteBRIDGE plating

SUMMARY:
The purpose of this combination retrospective and prospective post market study is to examine the short term safety and efficacy of the ROI-A® interbody fusion device with VerteBRIDGE® plates to treat single and two-level degenerative disc disease between L2 and S1, with a focus on fusion rates and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have degenerative disc disease (DDD) of the lumbar spine between L2 and S1
* Subjects may have up to a Grade 1 spondylolisthesis at the involved level(s)
* Subject must have the ROI-A® device at one level or at two contiguous levels between L2 and S1 only
* Subject should have had a minimum of 6 months non-surgical treatment prior to receiving the ROI-A® device
* Subject may have had NO MORE THAN two previous non-fusion surgeries to the lumbar spine at the same levels as the ROI-A®
* Subject must be at least 21 years of age at the time of surgery
* Subject must be willing to signed an informed consent document and return for a 12 month visit

Exclusion Criteria:

* Subject had more than Grade 1 spondylolisthesis at the operated level
* Subject is a prisoner.
* Subject was pregnant at the time of surgery.
* Subject had an active infection or sepsis at the time of surgery.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be drawn from community surgeon practices in which the subjects have already received the device and who meet the Inclusion/Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Operated Subjects
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Operated Subjects
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51
BMI (kg/mg^2) [Mean (Standard Deviation); unit: kg/mg^2] | 28.4 (4.6)
Current smoker [Count of Participants; unit: Participants] | 9
Previous Lumbar Spine Surgery [Count of Participants; unit: Participants] | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fusion
Description: Fusion was assessed utilizing both AP and flexion/extension radiographs. Fusion was noted when all three of the criteria were present: 1) presence of bridging bone as identified by radiography, 2)Less than 5 degrees of segmental motion on flexion/extension radiographs, and 3) Less than 3 mm of A/P translation on flexion/extension radiographs
Time Frame: 12 months after device implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Operated Subjects
Number analyzed (Participants) | 51
Participants | 50

2. Secondary Outcome: Mean Oswestry Disability Index
Description: The Oswestry Disability Index (ODI) is and index to quantify disability for low back pain. There are 50 possible points which are multiplied by 2 to arrive at a percentage score. Zero is equated with no disability and 100 is the maximum disability possible
Time Frame: 12 months after device implantation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Operated Subjects
Number analyzed (Participants) | 51
score on a scale | 28.9 (22.3)

ADVERSE EVENTS:
Time Frame: From enrollment through final follow up (12 month) visit
Description: An adverse event is defined as any change from baseline in a subject's condition during the clinical study. This includes events that are related to the device as well as events that are not related to the device.
Arm/Group | Operated Subjects
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 5/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operated Subjects (N=51)
Lower extremity neuropathy (Musculoskeletal and connective tissue disorders) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No